CLINICAL TRIAL: NCT04050111
Title: The Evaluation of Safety and Effectiveness of Intraarticular Administration of Autologous Stromal-Vascular Fraction of Adipose Tissue Cells for Treatment of Knee Joint Arthrosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Swiss Medica XXI Century S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SM-001
Record Dates: First submitted 2019-06-07; First posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Knee Osteoarthritis
Keywords: SVF; stromal-vascular fraction; Stem cell therapy
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SVF injection (Experimental): Subjects will undergo liposuction under local anesthesia. Lipoaspirate will be processed to isolate and concentrate stromal vascular fraction of cells (SVF). After SVF isolation autologous cells suspension will be injected intraarticularly into knee joint.
  Interventions:
  Procedure: Liposuction Other: SVF isolation Other: Intraarticular administration of autologous SVF
  Interventions: Biological: Stromal-vascular fraction

INTERVENTIONS:
Biological: Stromal-vascular fraction — Concentrate of stromal-vascular fraction of cells derived from autologous adipose tissue

SUMMARY:
Stromal vascular fraction of cells (SVF) will be extracted from lipoaspirate by enzymatic digestion. SVF will be administered in a single dose intraarticularly. All patients will receive cell therapy.This is a single arm study with no control.

DETAILED DESCRIPTION:
Patients with knee osteoarthritis will be subjected to abdominal liposuction under local anaesthesia. Harvested adipose tissue will be processed according to patent pending technology based on enzymatic digestion, washing and concentration of cell pellet in 5 ml of Hartmann's solution. Isolated SVF will be administered in a single dose into anterior part of knee joint cavity.

ELIGIBILITY:
Inclusion Criteria:

* Pain in the knee joint during more than a half day assessed by Visual Analog Pain Scale (score more than 40 mm)
* At least three of the following 6 criteria: 20-85 years of age, stiffness lasting less than 30 minutes, crepitus, bony tenderness, bony enlargement, no warmth to the touch
* Patient is able to walk without assistance
* Patient is familiar with Participant information sheet
* Patient signed informed consent form

Non-inclusion Criteria:

* Medical history of endoprosthetic knee replacement
* Medical history of lower extremity osteotomy
* Medical history of knee surgery (including arthroscopy) during preceding 1 year prior to enrollment
* Medical history of intraarticular injections during preceding 6 months prior to enrollment
* Secondary osteoarthritis of the knee joint: posttraumatic osteoarthritis (developed after clinically significant injury), intra-articular fractures, clinically significant varus or valgus deformities of lower limbs, septic arthritis, joint's inflammatory disorders, gout, advanced chondrocalcinosis, Paget's disease, ochronosis, acromegaly, hemochromatosis, Wilson's disease, primary synovial osteochondromatosis, osteonecrosis, hemophilia
* Patients prescribed for immunosuppressive treatment
* Medical history of systemic autoimmune and inflammatory diseases
* Significant weight loss (> 10% of body weight in the previous year) of unknown etiology
* Medical history of venous thromboembolism or estimated high risk of venous thromboembolism
* Patients prescribed for systemic corticosteroids or other medications treatment with proven impact on bone or cartilage tissue metabolism
* Clinically significant abnormalities in results of laboratory tests
* Any conditions limiting compliance (dementia, neuropsychiatric disease, drug and alcohol abuse etc.)
* Participation in other clinical trials (or administration of investigational drugs) during 3 months prior inclusion
* Patients with malignant tumors including postoperative period, patients receiving chemotherapy and/or radiotherapy.
* Patient's activated partial thromboplastin time exceeds normal levels more than 1,8 times
* Patients prescribed for anticoagulants treatment or patient received anticoagulants at least one hour prior liposuction
* Medical history of heterotopic ossifications
* Patients prescribed for glycoprotein inhibitors treatment

Exclusion Criteria:

* Patient's refusal from the further participation in trial
* Patient's refusal from compliance with the requirements of contraception during the participation in research
* Chronic kidney disease IV- V stages (creatinine clearance < 30 mL/min estimated by Cockcroft-Gault formula)
* Confirmed syphilis, HIV, hepatitis B or C infections

Dropout Criteria:

- Pregnancy

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-08-21 (Estimated); Primary Completion 2021-02-22 (Estimated); Study Completion 2021-08-22 (Estimated)

PRIMARY OUTCOMES:
Serious adverse events (SAEs) | 4 weeks after treatment
  Types, probability and severity of treatment emergent SAEs
Serious adverse reactions (SARs) | 4 weeks after treatment
  Types, probability and severity of treatment emergent SARs

SECONDARY OUTCOMES:
Quality of life monitoring-1 | Follow up to completion (up to 24 weeks after treatment)
  Quality of life estimated by validated questionnaire - the Short Form (36) Health Survey (SF-36).
  SF-36 is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  The eight sections are:
  * vitality
  * physical functioning
  * bodily pain
  * general health perceptions
  * physical role functioning
  * emotional role functioning
  * social role functioning
  * mental health
Quality of life monitoring-2 | Follow up to completion (up to 24 weeks after treatment)
  Quality of life estimated by validated questionnaire - Knee Injury and Osteoarthritis Outcome Score (KOOS).
  The KOOS is a patient reported joint-specific score, which assesses:
  * patient pain (9 items),
  * other symptoms (7 items),
  * function in daily living (17 items),
  * function in sport and recreation (5 items),
  * knee related quality of life (4 items).
  Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms.
Knee pain intensity monitoring | Follow up to completion (up to 24 weeks after treatment)
  Knee pain intensity assessed by Visual Analog Pain Scale (no pain=0; maximum pain=100 mm)
Changes in knee joint structure-1 | Follow up to completion (up to 24 weeks after treatment)
  Changes in knee joint structure assessed by ultrasonography (effusion, synovial thickening or hypertrophy, cartilage parameters, vascularity, Baker's cysts, osteophytes, tendon and ligament abnormalities, meniscal changes, bursitis, erosions and panniculitis)
Changes in knee joint structure-2 | Follow up to completion (up to 24 weeks after treatment)
  Changes in knee joint structure assessed by X-ray (joint space width, bone contour, presence of osteophytes and sclerosis)
Changes in knee joint structure-3 | Follow up to completion (up to 24 weeks after treatment)
  Changes in knee joint structure assessed by MRI (articular cartilage, osteophytes, bone marrow abnormality, meniscal integrity, synovial effusion/tissue, anterior and posterior cruciate ligaments, and medial and lateral collateral ligaments)
Changes in knee function | Follow up to completion (up to 24 weeks after treatment)
  Changes in knee function assessed by validated questionnaire: Knee Society Score (KSS).
  KSS consists of 4 separate sub-scales:
  * "Objective" Knee Score (seven items: 100 points),
  * Patient Satisfaction Score (five items: 40 points),
  * Patient Expectation Score (three items: 15 points),
  * Functional Activity Score (19 items: 100 points).
  Lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Sergey L Mikheev, MD, PhD, Principal Investigator — Head of Swiss Medica XXI Century S.A.; Ilya I Eremin, MD, PhD, Principal Investigator — Chief scientific officer of Swiss Medica XXI Century S.A.
Locations (2):
- Swiss Medica XXI Century S.A., Moscow, Russia
- IM Clinic, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No